CLINICAL TRIAL: NCT00885417
Title: The Efficacy of Sequential Therapy as Second Line Therapy for Refractory Helicobacter Pylori Infection - A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jyh-Ming Liou, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200901041M
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: H. Pylori Infection
Keywords: Helicobacter pylori; sequential therapy; levofloxacin; clarithromycin; rescue; salvage; treatment failure; For those who fail from one standard eradication therapy for H. pylori infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cravit-based sequential therapy (Experimental): Cravit-based sequential therapy Eligible patients will be treated with (esomeprazole 40mg bid +amoxicillin 1gm bid) for 5 days, followed by (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid ) for another 5 days
  Interventions: Drug: Cravit-based sequential therapy

INTERVENTIONS:
Drug: Cravit-based sequential therapy — Eligible patients will be treated with (esomeprazole 40mg bid +amoxicillin 1gm bid) for 5 days, followed by (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid ) for another 5 days

SUMMARY:
Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection could reduce the occurence or recurrence of these diseases. However, it was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy. About 15-30% of patient would fail from second line therapy and need to be rescued with third line therapy. The commonly used salvage regimens include:

1. Bismuth based quadruple therapy (combined with ranitidine or proton-pump inhibitor (PPI) plus two antibiotics)
2. Levofloxacin or moxifloxacin or rifabutin based triple therapy.

However, Bismuth is not available in many countries and the administration method is complex. Its usage is limited by the high pill number and low compliance rate. In recent years, the concept of sequential therapy has been advocated in the treatment of H. pylori infection. The regimen includes a PPI plus amoxicillin for five days, followed by a PPI plus clarithromycin and metronidazole for another five days. The eradication rate in the first line treatment of sequential therapy had been reported to be as high as 90%. More importantly, it has been demonstrated that the eradication rate among patients with clarithromycin-resistant strains could be as high as 89%.

Aims: Therefore, the investigators aim to assess the efficacy of levofloxacin-based sequential therapy as second line therapy for those who fail from one standard eradication therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged greater than 20 years who have persistent H. pylori infection after one treatment and are willing to receive second line rescue regimens, respectively, are considered eligible for enrollment.

Exclusion Criteria:

* Children and teenagers aged less than 20 years,
* History of gastrectomy,
* Gastric malignancy, including adenocarcinoma and lymphoma,
* Previous allergic reaction to antibiotics (amoxicillin, clarithromycin, levofloxacin) and prompt pump inhibitors (esomeprazole),
* Contraindication to treatment drugs,
* Pregnant or lactating women, OR
* Severe concurrent disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Eradication rate will be evaluated according to Intent-to-treat (ITT) and per-protocol (PP) analyses | 2009/4/20

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, Principal Investigator — Nationa Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan